CLINICAL TRIAL: NCT00562913
Title: Phase I Open-label, Non-randomized, Non-placebo Controlled Study to Determine the Safety, Pharmacokinetics, and Tumor Response Profile of Sorafenib as Continuous Dosing in Combination With Cyclophosphamide and Doxorubicin in Patients With Advanced, Refractory Solid Tumors
Brief Title: Phase I Study of Sorafenib Dosed Continuously With Cyclophosphamide and Doxorubicin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12347
Record Dates: First submitted 2007-11-21; First posted 2007-11-26 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Cancer
Keywords: Cancer; Sorafenib; Cyclophosphamide; Doxorubicin
MeSH Terms: conditions — Neoplasms | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Nexavar (Sorafenib, BAY43-9006)

INTERVENTIONS:
Drug: Nexavar (Sorafenib, BAY43-9006) — Cyclophosphamide plus 400 mg BID sorafenib and doxorubicin

SUMMARY:
Study to access the safety, levels of drug in the blood and tumor effects of sorafenib dosed daily combined with Cyclophosphamide and Doxorubicin in cancer patients

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Advanced histological or cytological documentation of cancer
* life-expectancy of at least 12 weeks
* able to swallow pills
* ECOG status of 0,1 or 2
* adequate bone marrow
* liver and renal function

Exclusion Criteria:

* > NYHA Class 2 CHF
* Serious myocardial dysfunction,
* or symptomatic coronary artery disease (MI more than 6 months prior to study entry is allowed)
* History of organ allograft
* uncontrolled hypertension
* renal dialysis
* Bleeding event/hemorrhage within 4 weeks of study treatment
* major surgery within 4 weeks of study treatment
* Previous exposure to doxorubicin or other anthracyclines exceeding a maximum lifetime cumulative dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine the pharmacokinetics and safety of cyclophosphamide when co-administered with 400 mg BID sorafenib and doxorubicin administered | 6 weeks

SECONDARY OUTCOMES:
To evaluate the tumor response to the combination of cyclophosphamide, doxorubicin and sorafenib | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Canada (2):
  - Edmonton, Alberta
  - Montreal, Quebec